CLINICAL TRIAL: NCT04475120
Title: Interventional Pilot Study to Assess the Use of Oral and Intra-nasal Liposomal Lactoferrin in COVID-19 Patients With Mild-to-Moderate Disease and in COVID-19 Asymptomatic Patients
Brief Title: Efficacy and Safety of Liposomal Lactoferrin in COVID-19 Patients With Mild-to-Moderate Disease and in COVID-19 Asymptomatic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Elena Campione, Associate Professor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4220
Record Dates: First submitted 2020-07-16; First posted 2020-07-17 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Liposomal Lacroferrin (Experimental): Thirty-two patients (14 hospitalised and 18 in home-based isolation) belonging to the first group received oral and intranasal liposomal bLf. BLf capsules for oral use containing 100 mg of bLf encapsulated in liposome while bLf nasal spray had about 8 mg/ml of bLf encapsulated in liposome. BLf, contained in both products, was tested by SDS-PAGE and silver nitrate staining and its purity was about 95%. The bLf iron saturation was about 5% as detected via optical spectroscopy at 468 nm based on an extinction coefficient of 0.54 (100% iron saturation, 1% solution). The scheduled dose treatment of liposomal bLf for oral use was 1gr per day for 30 days (10 capsules per day) in addition to the same formulation intranasally administered 3 times daily (a total of about 16 mg/nostril)
  Interventions: Drug: liposomal lactoferrin
- SOC therapy (Active Comparator): Thirty-two hospitalized patients belonging to the second group were only treated with SOC regimen according to the national guidelines at the time of the enrollment: lopinavir/ritonavir cps 200/50 mg, 2x2/day (alternatively darunavir 800 mg 1 cp/day+ritonavir 100 mg 1 cp/day or darunavir/cobicistat 800/150 mg 1 cp/day), chloroquine 500 mg, 1x2/day or hydroxychloroquine cp 200 mg, 1x2/day. SOC regimen lasted from 5 to 20 days, with timing to be established according to clinical course.
  Interventions: Drug: SOC therapy
- Home-based isolation (No Intervention): Twenty-eight patients, in home-based isolation, belonging to the third group did not receive any therapy.
- Healthy volunteers (No Intervention): A control group, comprising 32 healthy volunteers, did not receive any treatment or placebo.

INTERVENTIONS:
Drug: liposomal lactoferrin — oral and intra-nasal formulation
  Arms: Liposomal Lacroferrin
Drug: SOC therapy — oral administration
  Arms: SOC therapy

SUMMARY:
COVID-19 is considered an ongoing international global health problem which already caused 12 million confirmed cases. No specific effective treatment has been identified so far, and available supportive therapies are intended just to severe patients. Asymptomatic and mildly symptomatic patients remain a transmission reservoir, with possible evolution to the most severe disease form, without a clear treatment indication.

Lactoferrin (Lf) is a multifunctional glycoprotein, belonging to transferrin family, secreted by exocrine glands and neutrophils and present in all human secretion. The pleiotropic activity of Lf is mainly based on its four different functions: chelate two ferric iron per molecule, interact with anionic molecules, enter inside nucleus and modulate iron homeostasis. The ability to chelate two ferric ions per molecule is associated to the inhibition of reactive oxygen species formation as well as this sequestration of iron, pivotal for bacterial and viral replication, is at the basis of its antibacterial and antiviral activity. Moreover, Lf exerts its antiviral activity against the majority of the tested viruses by binding to heparan sulphate, while against few viruses by interacting with surface components of viral particles. The capability of Lf to exert antiviral activity, by binding to host cells or viral particles or both, strengthens the idea that this glycoprotein is "an important brick in the mucosal wall, effective against viral attacks". Lf was able to block the binding of the spike protein to host cells, indicating that Lf exerted its inhibitory function at the viral attachment stage. The current accepted model suggests that Lf could block viral entry by interacting with heparan sulfate proteoglycans (HSPGs), which mediate the transport of extracellular virus particles from the low affinity anchoring sites to the high affinity specific entry as ACE-2.

Investigators performed a prospective, interventional pilot study to assess the efficacy of liposomal lactoferrin in COVID-19 patients with mild-to moderate disease and in COVID-19 asymptomatic patients.

Secondary objectives evaluated the safety and tolerability of liposomal lactoferrin for oral and intra-nasal use.

DETAILED DESCRIPTION:
COVID-19 is considered an ongoing international global health problem which already caused 12 million confirmed cases. No specific effective treatment has been identified so far, and available supportive therapies are intended just to severe patients. Asymptomatic and mildly symptomatic patients remain a transmission reservoir, with possible evolution to the most severe disease form, without a clear treatment indication.

Lactoferrin (Lf) is a multifunctional glycoprotein, belonging to transferrin family, secreted by exocrine glands and neutrophils and present in all human secretion. The pleiotropic activity of Lf is mainly based on its four different functions: chelate two ferric iron per molecule, interact with anionic molecules, enter inside nucleus and modulate iron homeostasis. The ability to chelate two ferric ions per molecule is associated to the inhibition of reactive oxygen species formation as well as this sequestration of iron, pivotal for bacterial and viral replication, is at the basis of its antibacterial and antiviral activity.

Moreover, Lf exerts its antiviral activity against the majority of the tested viruses by binding to heparan sulphate, while against few viruses by interacting with surface components of viral particles. The capability of Lf to exert antiviral activity, by binding to host cells or viral particles or both, strengthens the idea that this glycoprotein is "an important brick in the mucosal wall, effective against viral attacks". Lf was able to block the binding of the spike protein to host cells, indicating that Lf exerted its inhibitory function at the viral attachment stage. The current accepted model suggests that Lf could block viral entry by interacting with heparan sulfate proteoglycans (HSPGs), which mediate the transport of extracellular virus particles from the low affinity anchoring sites to the high affinity specific entry as ACE-2.

Investigators performed a prospective, interventional, pilot study to assess the efficacy of liposomal lactoferrin in COVID-19 patients with mild-to moderate disease and in COVID-19 asymptomatic patients.

Secondary objectives evaluated the safety and tolerability of liposomal lactoferrin for oral and intra-nasal use.

Investigators conducted a parallel 3 group clinical trial to investigate the effect and tolerability of a liposomal bLf formulation as a supplementary nutraceutical agent in COVID19 patients. A total of 92 COVID19 patients, 25/92 asymptomatic and 67/92 mild-to-moderate, were recruited and divided into 3 groups according to the administered regimen: 32/92 COVID-19 patients, 14 hospitalised and 18 in home-based isolation, received oral and intranasal liposomal bLF supplement; 32 COVID-19 hospitalised patients were treated with hydroxychloroquine, azitromicin and lopinavir/darunavir as standard of care treatment (SOC); twenty eight COVID-19 patients, in home-based isolation did not take any medication against COVID-19. Furthermore, a group of 32 healthy subjects with negative COVID19 rRT-PCR was added as a control group for ancillary analysis.

Thirty-two patients (14 hospitalised and 18 in home-based isolation) belonging to the first group received oral and intranasal liposomal bLf. BLf capsules for oral use containing 100 mg of bLf encapsulated in liposome while bLf nasal spray had about 8 mg/ml of bLf encapsulated in liposome. BLf, contained in both products, was tested by SDS-PAGE and silver nitrate staining and its purity was about 95%. The bLf iron saturation was about 5% as detected via optical spectroscopy at 468 nm based on an extinction coefficient of 0.54 (100% iron saturation, 1% solution). The scheduled dose treatment of liposomal bLf for oral use was 1gr per day for 30 days (10 capsules per day) in addition to the same formulation intranasally administered 3 times daily (a total of about 16 mg/nostril) Thirty-two hospitalized patients belonging to the second group were only treated with SOC regimen according to the national guidelines at the time of the enrollment: lopinavir/ritonavir cps 200/50 mg, 2x2/day (alternatively darunavir 800 mg 1 cp/day+ritonavir 100 mg 1 cp/day or darunavir/cobicistat 800/150 mg 1 cp/day), chloroquine 500 mg, 1x2/day or hydroxychloroquine cp 200 mg, 1x2/day. SOC regimen lasted from 5 to 20 days, with timing to be established according to clinical course.

Twenty-eight patients, in home-based isolation, belonging to the third group did not receive any therapy.

A control group, comprising 32 healthy volunteers, did not receive any treatment or placebo.

Blood samples and clinical assessments were evaluated at baseline (T0), after 15 days (T1) and after 30 days (T2).

Eligible patients were over 20 years old, with a confirmed positivity to COVID-19 at the naso-oro-pharyngeal swab.

Exclusion criteria included pregnant and lactating women, patients taking nitric oxide and nitrates, patients with reported allergy to milk proteins, patients with a previous history of bronchial hyperactivity and patients with pre-existing respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients were over 20years old, with a confirmed positivity to COVID-19 at the oropharyngeal swab

Exclusion Criteria:

pregnant and lactating women, patients taking nitric oxide and nitrates, patients with reported allergy to milk proteins, patients with a previous history of bronchial hyperactivity and patients with pre-existing respiratory diseases. COVID-19 patients requiring intensive care or mechanical ventilation were excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Rate of viral clearance Time to viral clearance | 30 days
  time to naso-oro-pharingeal swab negativization

SECONDARY OUTCOMES:
Time to clinical improvement | 30 days
  time to improvement of clinical symptoms and blood parameters

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome Tor Vergata, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol